CLINICAL TRIAL: NCT01946542
Title: Acute Effects of Beet Juice Consumption on Exercise Capacity in Heart Failure
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Jason Allen, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Jason Allen, Ph.D., Assistant Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Pro00047311
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: exercise; heart failure; fatigue; physical endurance; functional food
MeSH Terms: conditions — Heart Failure; Motor Activity; Fatigue | interventions — Taste

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo drink, single dose, taste and color-matched to experimental drink
  Interventions: Other: placebo
- beet juice concentrate (Experimental): single dose of beet juice concentrate, roughly 70 mL
  Interventions: Drug: beet juice concentrate

INTERVENTIONS:
Drug: beet juice concentrate — single dose of beet juice concentrate, roughly 70 mL
  Arms: beet juice concentrate
Other: placebo
  Other Names: placebo drink, single dose, taste and color-matched to experimental drink
  Arms: placebo

SUMMARY:
The purpose of this project will be to determine whether consumption of beet juice concentrate prior to exercise may acutely improve exercise tolerance in patients with heart failure.

DETAILED DESCRIPTION:
Participants will complete up to four study visits. The first visit will involve completion of the informed consent process followed by a screening for study eligibility. The screening will consist of questionnaires pertaining to detailed medical history, diet, physical activity, and health-related quality of life (KCCQ). Anthropometric measures and a general health screening (including heart rate, resting blood pressure, and small blood (<15 mL) and urine samples will be collected). Volunteers meeting eligibility requirements will be scheduled for a screening maximal cardiopulmonary exercise test. Immediately prior to the exercise treadmill test, each subject will have a resting ECG and blood pressure to determine whether there are any abnormalities that would contraindicate exercise testing. Qualified subjects will then undergo a maximal cardiopulmonary exercise (CPX) test.

Following successful completion of the screening CPX test, volunteers meeting eligibility requirements will be scheduled for two testing visits, at least one week apart. At one visit, participants will consume a small cup of beet juice concentrate, and at the other, they will consume placebo. Treatment will be double-blinded and administered in random order.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) class II-III heart failure
* receiving optimal medical therapy
* sedentary

Exclusion Criteria:

* smoking
* changes in medication or major cardiovascular (CV) event or procedure within the previous 6 wk
* fixed rate pacemaker
* unstable angina
* other co-morbidities or limitations that preclude safe participation in the exercise testing
* plans for hospitalization or cardiac transplantation within the next 2 months
* type 1 diabetes
* refusal or inability to provide informed consent

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kraus, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 participants signed consent. 4 participants were screen failures. 2 participants were randomized.
Groups:
- Placebo First Then Beet Juice Concentrate: Testing visit 1: Participants are given a placebo drink, single dose. The placebo drink is taste and color-matched to the experimental drink.
  Testing visit 2: Participants are given a single dose of beet juice concentrate, roughly 70 mL.
- Beet Juice Concentrate First, Then Placebo: Testing visit 1: Participants are given a single dose of beet juice concentrate, roughly 70 mL.
  Testing Visit 2: Participants are given a placebo drink, single dose. The placebo drink is taste and color-matched to the experimental drink.
Period: Testing Visit 1
Arm/Group | Placebo First Then Beet Juice Concentrate | Beet Juice Concentrate First, Then Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Testing Visit 2
Arm/Group | Placebo First Then Beet Juice Concentrate | Beet Juice Concentrate First, Then Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First Then Beet Juice Concentrate | Beet Juice Concentrate First, Then Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1 | 0 | 1
  Black | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Exercise Tolerance
Description: treadmill time to exhaustion, cardiopulmonary exercise test
Time Frame: Testing Visit 1 (1-2 weeks from baseline) and Testing Visit 2 (2-3 weeks from baseline)
Population: Given that only one participant completed each arm of the study, we are unable to report outcomes as group means. To report the individual demographic, clinical, and/or physiological characteristics of these participants would present significant and unnecessary risk of loss of confidentially. Thus, no outcome data is reported.
Arm/Group | Placebo First Then Beet Juice Concentrate | Beet Juice Concentrate First, Then Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Vascular Function
Description: flow-mediated dilation (FMD)
Time Frame: Testing Visit 1 (1-2 weeks from baseline) and Testing Visit 2 (2-3 weeks from baseline)
Population: as for outcome 1
Arm/Group | Placebo First Then Beet Juice Concentrate | Beet Juice Concentrate First, Then Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: For the duration of study enrollment (Approximately 30 - 45 days)
Arm/Group | Placebo | Beet Juice Concentrate
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
The study was terminated due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No